CLINICAL TRIAL: NCT04969393
Title: Effects of High Intensity Laser on Mechanical and Physiological Findings in Pregnant Women With Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Effects of High Intensity Laser on Mechanical and Physiological Findings in Pregnant Women With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HILTPCTS2021
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Carpal Tunnel Syndrome; Pregnancy Related
Keywords: carpal tunnel syndrome; high intensity laser therapy; electrophysiology; pregnant women
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (High Intensity Laser therapy + Conventional Physical Therapy) (Experimental): Patients in group (A) received conventional physical therapy program along with HILT. Patients received pulsed Nd: YAG laser treatment, produced by EXAND MY 1064 nm Laser system, Mectronic Medicale, Italy. The apparatus provided pulsed emission (1064 nm), very high peak power (3 kW), a high level of fluency (energy density; 360-1780 mJ/cm2).
  Interventions: Device: High intensity laser therapy; Other: Conventional Physical Therapy
- Group B (Conventional Physical Therapy) (Active Comparator): Patients in this group received the conventional physical therapy program in the form of splinting, tendon and neural gliding exercises. Patients were instructed to wear a neutral custom volar splint at night and while performing strenuous activities during the day for 5 weeks.Also, the patients performed nerve-and tendon-gliding exercise under direct supervision of the therapist during the treatment sessions. Each exercise was repeated 10 times at each session and patients were encouraged to apply exercise 3-5 times per day for 5 weeks.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Device: High intensity laser therapy — Fifteen treatment sessions with pulsed Nd: YAG laser were applied to the subjects of the study group, three sessions per week, over 5 weeks in succession via EXAND MY 1064 nm Laser system, Mectronic Medicale, Italy. Patients in group (A) received HILT along with the conventional physical therapy program. The session involved 3 subphases: (1) The Initial phase "Analgesic phase", (2) In the intermediate phase "Trigger point phase"and (3)The final phase "Bio-stimulation phase" was applied for 6 minutes with a slow scanning in several parallel longitudinal lines.
  Other Names: High power laser therapy
  Arms: Group A (High Intensity Laser therapy + Conventional Physical Therapy)
Other: Conventional Physical Therapy — Fifteen treatment sessions that involved using a neutral custom volar splint alongside neural and tendon gliding exercises. the splint was used at night and while performing strenuous activities during the day for 5 weeks. While nerve and tendon gliding exercises was repeated 10 times at each session and patients were encouraged to apply exercise 3-5 times per day for 5 weeks.
  Other Names: Standard Physiotherapy

SUMMARY:
This study will propose a novel approach to treat pregnant women with mild to moderate carpal tunnel syndrome (CTS) using the recently introduced High intensity laser therapy with its deep penetration and high-power characteristics. It's hopeful that the results of this study can fill the gap of knowledge surrounding the conservative treatment options for CTS in order to help patients restore their nerve function properly and promote new ways of addressing CTS.

ELIGIBILITY:
Inclusion Criteria:

(1) Pregnant women with mild to moderate CTS diagnosed by a physician according to the American Association of Electrodiagnostic recent guidelines [18] (2) The age ranged between 20 to 40 years (3) Had positive clinical provocative tests for the CTS (Tinel test and Phalen test) and (5) Had a history of pain, paresthesia or numbness in the median nerve distribution, nocturnal pain, and night waking

Exclusion Criteria:

Patients were excluded from the study if they had cervical disc prolapse, cervical spondylosis, thoracic outlet syndrome, diabetes, gestational diabetes, cardiovascular disorders and hypertension. Patients who had carpal tunnel release surgery and patients who were diagnosed with CTS before pregnancy were also excluded from the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Distal latency of median nerve sensory distal latency | Baseline and after 5 Weeks
  The Median sensory nerve (SNDL) distal latency was measured according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines with a Neuropack S1 MEB-9004 Nihon Koden (Japan). All measurements were performed in a room with the temperature kept at 25C.
Changes in Distal latency of median nerve motor distal latency | Baseline and after 5 Weeks
  The Median motor nerve (MNDL) distal latency was measured according to the American Association of Electrodiagnostic Medicine (AAEM) guidelines with a Neuropack S1 MEB-9004 Nihon Koden (Japan). All measurements were performed in a room with the temperature kept at 25C.

SECONDARY OUTCOMES:
Changes in hand grip strength | Baseline and after 5 Weeks
  The hand grip strength (measured in Kilograms) was evaluated by the same investigator. Grip strength was tested by using Jamar hand held dynamometer following the American Society of Hand Therapists guidelines. The patient's arm was positioned with the shoulder adducted and neutrally rotated, the elbow was flexed at 90, the forearm and wrist were neutrally positioned while the participant was sitting. Patients were instructed to squeeze the handle as hard as they could, do maximal grip contraction for 2-5 s.
Changes in numeric pain rating scale (NPRS) | Baseline and after 5 Weeks
  An 11-point Numerical Pain Rating Scale (NPRS; 0 = no pain, 10 = maximum pain) was used to assess the patients' levels of hand pain pre and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer F Hanafy, Ph.D, Study Chair — Cairo University; Radwa M Yehia, Ph.D, Study Director — Faculty of Physical Therapy, October 6 University
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial and after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 Months after study publication
Access Criteria: Email: mohamed.magdy.pt@o6u.edu.eg